CLINICAL TRIAL: NCT02994264
Title: A Retrospective Cohort Study to Assess Adjuvant Concurrent Chemoradiation (CCRT) Compared to Adjuvant Radiation Therapy (RT) in the Treatment of Grade 2 and 3 Extremity Soft Tissue Sarcomas
Brief Title: A Study to Compare Adjuvant Concurrent Chemoradiation (CCRT) to Adjuvant Radiation Therapy (RT) in Grade 2 and 3 Extremity Soft Tissue Sarcomas
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: ICL_2015_0002
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Sarcoma,Soft Tissue
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Radiation: adjuvant concurrent chemoradiation

SUMMARY:
The aim of the study is to retrospectively evaluate the outcome of adjuvant concurrent chemoradiation delivered to patients with high grade non-metastatic soft tissue sarcomas of the extremities at the investigators institution paired with patients treated by adjuvant radiation therapy

ELIGIBILITY:
Inclusion Criteria:

* All patients consecutive enrolled from 1990 to 2004 with soft tissue sarcomas located either in the limbs or girdles, superficial or deep, grade 2 or 3 (FNCLCC), who were first treated with radical conservative surgery and adjuvant RT atto a minimum biologically equivalent dose of 45 Gy, with or without concurrent adjuvant chemotherapy.

Exclusion Criteria:

* A patient record captured outside the time frame from 1990 to 2004 with trunk, retro-peritoneum, and head and neck localisations, grade 1 histology and, PS≥3, were excluded as well as and those plus patients who had received neoadjuvant treatment. Differentiated liposarcomas, dermatofibrosarcomas protuberans, extraskeletal Ewing's sarcomas, primitive neuroectodermal tumors and osteosarcomas were also excluded due to specific treatment strategies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients records would be extracted from the electronic health record system of Institut de Cancérologie de Lorraine
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
overall survival | 60 months